CLINICAL TRIAL: NCT05946148
Title: Effect of Dulaglutide vs Empagliflozin on Non-alcoholic Fatty Liver Disease of Patients With Type 2 Diabetes Mellitus
Brief Title: Novel Antidiabetic Medications and Their Effect on Liver Steatosis (NAMELS-18)
Acronym: NAMELS-18
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Alexandra Hospital, Athens, Greece (Other); Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, KOULLIAS EMMANOUIL, INTERNIST, National and Kapodistrian University of Athens
Other Study IDs: SC12/16-6-2016
Record Dates: First submitted 2023-07-05; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Liver Steatosis
Keywords: Empagliflozin; Dulaglutide; Liver Steatosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — empagliflozin; dulaglutide; Fumigant 93; Tin Fluorides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 vials of serum taken at each patient visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Empagliflozin group: Oral Empagliflozin 10mg daily, as add-on to their previous treatment regimen.
  Interventions: Drug: Empagliflozin
- Dulaglutide group: Subcutaneous Dulaglutide 1.5mg weekly, as add-on to their previous treatment regimen.
  Interventions: Drug: Dulaglutide
- Control group: Optimal anti-diabetic treatment (apart from agents of the GLP1-ras or SGLT2-is families), targeting glycemic control.
  Interventions: Drug: Control Rx

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin 10mg daily, as add-on to previous treatment regimen.
  Other Names: E
  Groups: Empagliflozin group
Drug: Dulaglutide — Dulaglutide 1.5mg weekly, as add-on to previous treatment regimen
  Other Names: D
  Groups: Dulaglutide group
Drug: Control Rx — Optimal anti-diabetic treatment excluding agents of the GLP1-ras or SGLT2-is families.
  Other Names: C
  Groups: Control group

SUMMARY:
The goal of this clinical study is to compare the therapeutic effect of Dulaglutide and Empagliflozin in patients with Diabetes Mellitus type 2 and Non-Alcoholic Fatty Liver Disease. The main question it aims to answer is: Is there a beneficial effect regarding liver steatosis in patients receiving either of these 2 medications and which is more effective? Patients will undergo shearwave elastography, magnetic resonance imaging, and ultrasound. Furthermore, calculation of the Fatty Liver Index (FLI), the Fibrosis-4 Index (FIB-4), as well as the Aspartate Aminotransferase to Platelet ratio Index (APRI) and the NAFLD Fibrosis Score (NFS) will be performed.

Researchers will compare 3 groups:

Group 1 will receive oral Empagliflozin, as add-on to their previous treatment regimen, for 52 weeks.

Group 2 will receive subcutaneous Dulaglutide, as add-on to their previous treatment regimen, for 52 weeks.

Group 3 will receive other optimal antidiabetic treatment (apart from agents of the GLP1-ras or SGLT2-is families) for 52 weeks.

DETAILED DESCRIPTION:
Rationale:

NAFLD is the most common chronic liver disease worldwide. Presently, relative clinical guidelines focus on weight loss through apporopriate diet and lifestyle. The Glucagon-Like Peptide 1 receptor agonists and the Sodium-Glucose Co-transporter 2 inhibitors constitute novel agents that seem to exert beneficial effects beyond glycemic control. Dulaglutide will be used from the GLP1-ras family and Empagliflozin from the SGLT2-is family.

Research question:

Is the use of Empagliflozin or Dulaglutide effective in improving liver fat fraction in patients with type 2 diabetes mellitus and NAFLD? Which is more beneficial?

Hypothesis:

The investigators hypothesize that both Dulaglutide and Empagliflozin have a role in treating patients with DM2 and NAFLD.

Aim of the study:

To compare the effect of Dulaglutide and Empagliflozin in liver fat fraction of diabetic patients after a year of treatment.

Objectives:

Assess liver steatosis change in patients. Determine percentage of those with >30% liver fat concentration reduction.

Compare Empagliflozin group with Dulaglutide group and Control group. Evaluate the impact of the medications used on glycemic control, weight loss, liver enzymes, lipids and the Fatty Liver Index (FLI), the Fibrosis-4 Index (FIB-4), as well as the Aspartate Aminotransferase to Platelet ratio Index (APRI) and the NAFLD Fibrosis Score (NFS).

Material and methods:

Site of study:

This study will be conducted in the 2nd Department of Internal Medicine of Hippocration General Hospital, and the Therapeutic Department of General Hospital "Alexandra", Athens, Greece.

Type of study:

This is a prospective open-label observational study.

Subjects allocation:

Group 1: patients will receive oral Empagliflozin, as add-on to their previous treatment regimen, for 52 weeks.

Group 2: patients will receive subcutaneous Dulaglutide, as add-on to their previous treatment regimen, for 52 weeks.

Group 3: patients will receive other optimal antidiabetic treatment (apart from agents of the GLP1-ras or SGLT2-is families) for 52 weeks.

Patients receiving Pioglitazone were not included in the study.

Steps of performance and techniques:

Medical history and complete physical examination. Informed consent. Calculation of BMI, measurement of waist and hip circumference. Blood tests including: Liver function tests, Complete blood count, Urea and Creatinine, Lipid profile (total cholesterol, triglycerides, LDL, HDL), fasting plasma glucose and HbA1c.

Abdominal ultrasound, Magnetic Resonance Imaging-Proton Density Fat Fraction, Shearwave Elastography.

Calculation of the Fatty Liver Index (FLI), the Fibrosis-4 Index (FIB-4), as well as the Aspartate Aminotransferase to Platelet ratio Index (APRI) and the NAFLD Fibrosis Score (NFS).

Assessment of changes between date of entry in the study and 52 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

Presence of diabetes mellitus type 2 and non-alcoholic fatty liver Stable anti-diabetic treatment regimen for the past 6 months

Exclusion Criteria:

Recent (last 5 years) medical history of cancer, pancreatitis, viral hepatitis or any other cause of liver disease (alcohol abuse, autoimmune hepatitis, hemochromatosis, heart failure etc.) Recent alteration (<6 months) of anti-diabetic regimen. Already established treatment with GLP1-ras or SGLT2-is prior to screening. Treatment with Pioglitazone. Corticotherapy administration. Pregnant or planning for pregnancy.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian, 25-75 years old, diagnosed with type 2 diabetes mellitus and fatty liver.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Liver Fat Fraction reduction | 52 weeks
  Change of Liver Fat Fraction as calculated by MRI-PDFF
>30% Liver Fat Fraction reduction | 52 weeks
  Percentage of each group's participants that achieves >30% Liver Fat Fraction reduction

SECONDARY OUTCOMES:
HbA1c change | 52 weeks
  Evaluation of HbA1c change in each group
Body Mass Index change | 52 weeks
  Evaluation of Body Mass Index change in each group
Fatty Liver Index (FLI) | 52 weeks
  Evaluation of FLI change in each group.
Fibrosis-4 Index (FIB-4) | 52 weeks
  Evaluation of FIB-4 change in each group.
Aspartate Aminotransferase to Platelet ratio Index (APRI) | 52 weeks
  Evaluation of APRI change in each group.
NAFLD Fibrosis Score (NFS) | 52 weeks
  Evaluation of NFS change in each group.
Shearwave Elastography (SWE) | 52 weeks
  Evaluation of SWE change in each group.

CONTACTS AND LOCATIONS:
Overall Officials: JOHN KOSKINAS, PROFESSOR, Study Chair — National and Kapodistrian University of Athens; ANASTASIA THANOPOULOU, AS PROFESSOR, Study Director — National and Kapodistrian University of Athens; MELANIE DEUTSCH, AS PROFESSOR, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- "Hippocration" General Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after analysis is completed and study results have been published. Expected to happen in 1st Semester of 2024. It will include participants' results of imaging and laboratory examinations in excel files.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: Upon request